CLINICAL TRIAL: NCT06267859
Title: Based on Medical Statistical Analysis and Screening (Dispensary) Examination, Identification of the Most Common Somatic and Congenital Diseases in Children, With the Further Development of More Effective Methods of Treatment and Recovery
Brief Title: Development of Methods for Effective Treatment and Improvement of Common Somatic Diseases in Children
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tashkent State Medical University (Tashkent Pediatric Medical Institute), Uzbekistan (Other)
Responsible Party: Principal Investigator, Turdieva Shokhida Tolkunovna, MD, Doctor of Medical Sciences, Professor, Tashkent State Medical University (Tashkent Pediatric Medical Institute), Uzbekistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: No. 2 of 2023/11/7
Record Dates: First submitted 2023-12-20; First posted 2024-02-20 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Diseases; Congenital Heart Defects
Keywords: children; adolescents; heart diseases; lung diseases; congenital malformations
MeSH Terms: conditions — Respiratory Tract Diseases; Heart Defects, Congenital; Heart Diseases; Lung Diseases; Congenital Abnormalities

STUDY DESIGN:
Intervention Model Description: identification of children from the group of "frequently ill children"
Who Masked: Participant
Masking Description: working with children from the "frequently ill children" group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- First stage (No Intervention): Study of children from the group of "frequently ill children", and with congenital diseases, collection of anamnesis, their examination, clinical and laboratory examination. Purpose: to identify the most frequently encountered group of diseases among children.
- Second stage (No Intervention): Study the effectiveness of treatment according to approved treatment standards
- third stage (No Intervention): Based on the research results, develop your treatment tactics. It is approved by the Ethics Committee for working with patients.
- fourth stage (Experimental): Use your treatment tactics among a group of patients. Study the effectiveness of the proposed therapy and rehabilitation methods.
  Interventions: Combination Product: The use of a combination of microelements and vitamins against the background of physiotherapy
- fifth stage (No Intervention): Based on the research data, clinical recommendations for doctors will be developed.

INTERVENTIONS:
Combination Product: The use of a combination of microelements and vitamins against the background of physiotherapy — If necessary, necessary microelements and vitamins will be added to the treatment process. At the same time, physiotherapeutic procedures will be added at the rehabilitation stage.
  Arms: fourth stage

SUMMARY:
The goal of the clinical study is to clarify the course of common congenital, infectious, and non-infectious diseases in children living in Uzbekistan, and to develop methods for their treatment and rehabilitation.

The main questions it aims to answer:

* Analysis of common congenital diseases among children;
* Analysis of commonly diagnosed bronchopulmonary and cardiovascular diseases among children;
* Based on the results of the primary research, common diseases among children will be identified;
* Analysis of existing treatment methods and their effectiveness;
* Development of modern methods of treatment and rehabilitation of children.

DETAILED DESCRIPTION:
Children's health is a priority in modern medicine. Some childhood diseases are most often encountered in the practice of pediatricians and family doctors. Children with these diseases need early diagnosis, treatment, and rehabilitation.

Patient selection criteria are:

* children from birth to 15 years;
* children permanently residing in the territory where the clinical examination is carried out;
* children included in the group of "frequently ill children";
* patients without severe chronic diseases.

Exclusion criteria:

* Teenagers over 15 years old;
* Patients with severe neurological and mental diseases;
* Patients with endocrinological diseases;
* Patients with long-term chronic somatic diseases;
* Children without genetic pathologies.

Clinical research methods:

* Collection of anamnestic data;
* General examination of patients (auscultation, palpation, percussion);
* If necessary: consultation with a geneticist and pediatric doctors of various specialties (cardiologist, surgeon, urologist, nephrologist, otolaryngologist, pulmonologist, immunologist, allergist)
* Standard laboratory tests (general analysis of blood, urine, feces);
* Standard biochemical studies (microelements of blood and enzymes in venous blood);
* Instrumental studies: chest X-ray, ultrasound examination of internal organs (chest and abdominal organs), computed tomography (chest and abdominal organs);
* Study of immunological status (cellular immunity, according to standard methods); Immunological research methods - flow cytometry, mIU/mL: immunogram - CD3, CD3/4, CD3/8, CD19, CD16/56, CD3/16/56, CD3/HLA-; and others;
* Study of antioxidant status (TAS, using the PSR method, mmol/L);
* Assessing the quality of life of patients (methods: PedsQLtm 4.0; HBSC, indicator: total score on the screening survey).

ELIGIBILITY:
Inclusion Criteria:

* children from birth to 15 years;
* children permanently residing in the territory where the clinical examination is carried out;
* children included in the group of "frequently ill children";
* patients without severe chronic diseases.

Exclusion Criteria:

* Teenagers over 15 years old;
* Patients with severe neurological and mental diseases;
* Patients with endocrinological diseases;
* Patients with long-term chronic somatic diseases;
* Children without genetic pathologies.

Ages: 3 Days to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2033-12-30 (Estimated); Study Completion 2034-01-30 (Estimated)

PRIMARY OUTCOMES:
Working with archival documentation. | one year
  Medical and statistical analysis of data from children's medical institutions is carried out to identify common somatic diseases in children from birth to 15 years old associated with impaired immunity.
  Evaluation criterion:
  * medical archival documentation of children's clinics in the region;
  * statistical analysis of archival documentation on the morbidity of children (acute respiratory: acute bronchitis and acute pneumonia; cardiovascular diseases: congenital heart disease, congenital and acquired carditis).
Formation of a group of patients to study immunity and the antioxidant system in venous blood. | one year
  Objective: Preparations for a clinical trial are underway.
  Work in progress:
  * 400 children with diseases of the bronchopulmonary system and congenital heart defects will be selected;
  * preparation and submission to the Ethics Committee under the Ministry of Health of Uzbekistan of all necessary documentation for the planned clinical trial among children;
  Evaluation criterion:
  - The percentage of detection of acute bronchopulmonary and congenital heart defects in the region of residence (results of medical statistics).
Clinical scientific research. | five years.
  A clinical study of sick children (acute respiratory: acute bronchitis and acute pneumonia; cardiovascular diseases: congenital heart disease, congenital and acquired carditis) is being conducted to determine the presence of immunological and antioxidant blood parameters.
  Work in progress:
  * Screening medical examination of children (objective examination, general blood test - ELISA method);
  * Examination of venous blood for indicators of immune status (extended immunogram: CD3, CD3/4, CD3/8, CD19, and others), method: flow cytometry of venous blood, mIU/mL;
  * the study of antioxidant status in sick children (Total antioxidant status, method: venous blood PCR, mmol/L);
  * publication of the research results.
  Evaluation criterion:
  * opinion of reviewers and experts in this field (comparison of the results obtained by other scientists - immunological and antioxidant research)
  * changes in immune and antioxidant status indicators in sick children to healthy peers.
Clinical trial evaluation. | three years
  The development and implementation of clinical recommendations for practicing pediatricians, pediatric pulmonologists, and cardiologists on improving children's health with acute respiratory (acute bronchitis, pneumonia) and cardiovascular (CHD, congenital and acquired carditis) diseases.
  Work in progress:
  * development and implementation of clinical recommendations for pediatricians, pediatric pulmonologists, and cardiologists;
  * assessment of the effectiveness of clinical recommendations based on repeated laboratory tests (immunological (flow cytometry, mIU/mL) and TAS (PCR, mmol/L)), after six months of implementation of the recommendations.
  Evaluation criterion:
  * opinion of reviewers and experts - review;
  * assessing the quality of life of patients (methods: PedsQLtm 4.0; HBSC), indicator: total score on the screening survey;
  * number of recurrent illnesses and complications, indicator: the number of patients as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Shokhida T Turdieva, D.Sc., Principal Investigator — Tashkent State Medical University (Tashkent Pediatric Medical Institute), Uzbekistan
Locations (1):
- Turdieva Shokhida Tolkunovna, Tashkent, Yunus-obad District, Uzbekistan

IPD SHARING:
Plan to Share IPD: Yes
This clinical study aims to discover the course of common congenital, infectious, and non-infectious diseases among children living in Uzbekistan, to develop methods for their treatment and improvement. Several separate clinical studies by young scientists will be combined.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2034/01/30
Access Criteria: Researchers at the Tashkent Pediatric Medical Institute.